CLINICAL TRIAL: NCT06849531
Title: Evaluation of the Relationship Between Foot Biomechanics and Lower Extremity Muscle Mechanics, Strength and Balance
Brief Title: Foot Biomechanics and Lower Extremity Muscle Mechanics
Status: Not yet recruiting | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Derya Azim, Assistant Professor, Bandırma Onyedi Eylül University
Other Study IDs: 2024-164
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Balance; Lower Extremity; Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Foot Biomechanics and Lower Extremity Muscle Analysis — Focus on Foot Biomechanics

SUMMARY:
This study is designed to investigate the relationship between foot biomechanics, balance, lower extremity muscle mechanical properties, and vertical jump in young adults. The aim is to highlight the correlations between foot biomechanics and the other parameters, as well as potential outcomes (if any).

DETAILED DESCRIPTION:
This study is designed to investigate the relationship between foot biomechanics, balance, lower extremity muscle mechanical properties, and vertical jump in young adults. The independent variables of the study include participants' age, height, weight, calcaneotibial angle, navicular drop test, foot lengths, smoking/alcohol habits, socioeconomic status, and exercise habits. The dependent variables are the results from the Korebalance balance test, Flamingo balance test, vertical jump test, and Myoton-Pro assessment. The study aims to highlight the correlations between foot biomechanics and the other parameters, as well as potential outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study
* Aged between 18 and 25 years
* No regular exercise habits

Exclusion Criteria:

* Having a physical disability that prevents participation in the study (e.g., use of a wheelchair, walker, and/or crutches, etc.)
* Having conditions that directly affect balance, such as vertigo or multiple sclerosis (MS)
* Having a neurological disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young adults
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-03-13 (Estimated); Primary Completion 2025-05-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
muscle mechanics | Single assessment at baseline
  The mechanical properties of the relevant muscle were measured at its midpoint using the MyotonPRO device, and the first three values were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Azim, Principal Investigator — Bandırma Onyedi Eylül University
Locations (1):
- Bandırma Onyedi Eylul University, Balıkesir, Bandırma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided